CLINICAL TRIAL: NCT07155707
Title: Phase II: Engagement and Clinical Impact of the Teleo Virtual Therapy Platform in Clinical Settings
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); MainSquare Co. (dba 'Teleo') (Unknown)
Responsible Party: Principal Investigator, David Hong, Associate Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 80119; R42MH136878 (NIH)
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Mood Disorders
Keywords: Teletherapy; Therapeutic Engagement; Anxiety; Depression; Youth Mental Health; Digital Mental Health
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teleo (Experimental): Participants in this arm will undergo therapy for 12 sessions using the Teleo virtual therapy video platform. Sessions will be recorded and questionnaires and clinical data will be measured.
  Interventions: Other: Teleo
- Standard Videoconferencing (Active Comparator): Participants in this group will undergo therapy for 12 sessions using standard video platforms (e.g. Zoom or Microsoft Teams). Sessions will be recorded and questionnaires and clinical data will be measured.
  Interventions: Other: Standard Videoconferencing

INTERVENTIONS:
Other: Teleo — Therapist-led psychotherapy sessions implemented within the Teleo virtual therapy platform.
  Arms: Teleo
Other: Standard Videoconferencing — Therapist-led psychotherapy sessions implemented in standard (non-Teleo) video platform.
  Arms: Standard Videoconferencing

SUMMARY:
This Phase II trial will examine engagement in telehealth for children undergoing psychotherapy. Specifically, the trial will examine patient engagement in Teleo, a virtual therapy platform specifically designed for psychotherapy with youth, as compared to standard video conferencing.

DETAILED DESCRIPTION:
This study aims to examine the impact of tailored telehealth psychotherapy environments on clinical outcomes in the context of pediatric mental health treatment. Researchers will conduct a full-scale RCT with 156 families to assess how Teleo compares to standard video conferencing (e.g., Zoom) on a range of clinical metrics, including cancellation/no-show rates, clinician satisfaction, duration of treatment, need for medication, and symptoms of anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a mood and/or anxiety disorder
* Have proficiency to participate in psychotherapy in English
* Scheduled to begin therapy at one of the study sites
* RCADS score > 65

Exclusion Criteria:

- Comorbid diagnosis of intellectual disability, autism spectrum disorder, psychotic disorders, high-risk suicidal behaviors requiring immediate hospitalization, substance use disorders, or other physical or mental condition that would prohibit them from engaging in telehealth settings.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Child Involvement Rating Scale (CIRS) | Week 1
  Observational coding questionnaire designed to assess child engagement in therapy. Consists of 6 items (4 positively-framed, 2 negatively-framed), each on a 0-5 scale. To calculate a summary score, the two negatively-framed items are reverse scored and scores on all six items are averaged. Summary scores range from 0-5, with higher scores representing greater child engagement in therapy.

SECONDARY OUTCOMES:
My Thoughts About Therapy Scale - Caregiver (MTT-CG) | Weeks 1, 6 and 12
  Caregivers will complete the MTT-GC questionnaire to measure their child's engagement in psychotherapy across dimensions of the REACH client engagement framework - Relationship, Expectancy, Attendance, Clarity, and Homework. Scores range from 0-105, higher scores indicate 'better' outcome.
My Thoughts About Therapy Scale - Youth (MTT-Y) | Weeks 1, 6 and 12
  Youth will complete questionnaires to measure self-reported engagement in psychotherapy across dimensions of the REACH client engagement framework - Relationship, Expectancy, Attendance, Clarity, and Homework. Scores range from 0-105, higher scores indicate 'better' outcome.
Revised Children's Anxiety and Depression Scale (RCADS) | Baseline, Week 4, Week 12
  Caregivers will complete questionnaire to assess child participants' symptoms of anxiety and mood disorders across six dimensions: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). Standardized T-scores will be calculated for each subscale and for the overall scale. T-scores range from 30-90, with lower scores representing better outcomes.
Rate of therapy session cancellations, no-shows, and treatment dropout | Weeks 1-12
  Participants' electronic health records (EHR) will be used to track session cancellations, no-shows, and treatment dropout.
Rate of clinician attrition | Weeks 1-12
  Clinician attrition rates will be assessed via electronic health records (EHR).
Long-Term Cost of Care | 1 year post-enrollment
  Treatment duration and medication use will be assessed over 1 year following participants' enrollment in the study, and used to calculate differences in average long-term cost of care between the study arms.

CONTACTS AND LOCATIONS:
Overall Officials: David S Hong, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Ohana Center for Child and Adolescent Behavioral Health, Monterey, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No